CLINICAL TRIAL: NCT03952806
Title: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of BHV-3241 in Subjects With Multiple System Atrophy (M-STAR Study)
Brief Title: Study of BHV-3241 in Participants With Multiple System Atrophy
Acronym: M-STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3241-301
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Results first posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy (MSA)
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind to Sponsor, Investigator and Subject
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verdiperstat (Experimental): Participants received verdiperstat 300 mg tablet orally once daily for 1 week, followed by 300 mg twice daily for 1 week, and then 600 mg twice daily for the remaining 46 weeks of the double-blind phase.
  Participants who completed the double-blind phase were offered the opportunity to enroll in an open-label extension (OLE) phase to continue verdiperstat 600 mg twice daily for 48 weeks.
  Interventions: Drug: Verdiperstat
- Placebo (Placebo Comparator): Participants received placebo matching with verdiperstat for 48 weeks. Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to receive verdiperstat 600 mg tablet orally twice daily for 48 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Verdiperstat — 300mg 2 oral tablets, twice daily
  Arms: Verdiperstat
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of verdiperstat (BHV-3241) versus placebo in participants with Multiple System Atrophy

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable or possible MSA according to consensus clinical criteria (Gilman et al 2008), including participants with MSA of either subtype (MSA-P or MSA-C).
2. Able to ambulate without the assistance of another person, defined as the ability to take at least 10 steps. Use of assistive devices (e.g., walker or cane) is allowed.
3. Anticipated survival of at least 3 years at the time of Screening, as judged by the Investigator.

Exclusion Criteria:

1. Any condition that would interfere with the participant's ability to comply with study instructions, place the participant at unacceptable risk, and/or confound the interpretation of safety or efficacy data from the study, as judged by the Investigator.
2. Diagnosis of neurological disorders, other than MSA.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (29):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UC San Diego Department of Neurosciences, La Jolla, California
  - UCLA Medical Center / Neurological Services, Los Angeles, California
  - Stanford University, Palo Alto, California
  - UCSF Memory and Aging Center, San Francisco, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Albany Medical College, Albany, New York
  - NYU School of Medicine, NYU Dysautonomia Center, New York, New York
  - Columbia University Medical Center, Neurological Institute, New York, New York
  - Pennsylvania State University Hershey Medical Center, Hershey, Pennsylvania
  - Parkinson's Disease and Movement Disorders Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kerwin Research Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Swedish Medical Center, Seattle, Washington
- Austria (2):
  - Confraternitaet Privatklinik Josefstadt in Wien, Vienna, Vienna
  - University Clinic Innsbruck, Innsbruck
- France (5):
  - CHU de Bordeaux, Service de Neurologie, Bordeaux
  - CHU - Hospital de la Timone, Marseille
  - Unité d'investigation clinique de Neurologie Rez-de-jardin, Bloc Hopital CHU Pontchaillou, Rennes
  - Hopitaux Universitaire de Strasbourg-Centre de References des Maladies Autoimmunes, Strasbourg
  - CHU Purpan, Toulouse
- Germany (9):
  - University Hospital of Liepzig, Leipzig, Saxony
  - St. Josef - Hospital Bochum, Kardiologische Studienambulanz, Bochum
  - Deutsches Zentrum für Neurodegenerative Erkrankungen (DZNE), Bonn
  - University Hospital Duesseldorf, Düsseldorf
  - CRC Core Facility Medizinische Hochschule Hannover (MHH), Hanover
  - Paracelsus-Elena-Klinik, Kassel
  - Klinik für Neurologie - UKSH - Campus Kiel, Kiel
  - Universitaetsklinikum Giessen und Marburg GmbH - Parkinson-Studienzentrum, Klinik für Neurologie, Marburg
  - Universitaetsklinikum Muenster, Münster
- Italy (2):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico di Milano, Milan, Milan
  - A.O.U. San Giovanni di Dio e Ruggi d'Aragona, Salerno
- The Newcastle upon Tyne Hospitals NHS Foundation Trust - Campus for Ageing and Vitality (NGH), Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Schmahmann JD, Pierce S, MacMore J, L'Italien GJ. Development and Validation of a Patient-Reported Outcome Measure of Ataxia. Mov Disord. 2021 Oct;36(10):2367-2377. doi: 10.1002/mds.28670. Epub 2021 Jun 11. PMID 34115419

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, randomized, double-blind, placebo-controlled study was conducted in participants with multiple system atrophy (MSA) at 48 centers in the US and EU between 29-Jul-2019 and 29-Jul-2021.
Pre-assignment Details: A total of 421 participants were enrolled, of which 336 participants were randomized in a 1:1: ratio to receive verdiperstat or placebo. 85 participants were not randomized due to withdrawal of consent, adverse events, failed inclusion/exclusion criteria, or other reasons.
Groups:
- Verdiperstat: Randomization phase (Randomization through Week 48): Participants received verdiperstat 300 milligrams (mg) tablet orally once daily for 1 week, followed by 300 mg twice daily for 1 week, and then 600 mg twice daily for the remaining 46 weeks of the double-blind phase.
  Open-label extension (OLE) phase (48 weeks): Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to continue verdiperstat 600 mg orally twice daily for 48 weeks.
- Placebo: Randomization phase (Randomization through Week 48): Participants received placebo matching with verdiperstat for 48 weeks.
  OLE phase (48 weeks): Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to receive verdiperstat 600 mg tablet orally twice daily for 48 weeks.
Period: Randomization Phase (Weeks 1 Through 48)
Arm/Group | Verdiperstat | Placebo
Started | 168 | 168
Completed | 127 | 146
Not Completed | 41 | 22
Not completed — Adverse Event | 26 | 15
Not completed — Disease progression | 5 | 0
Not completed — Participant request | 5 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Other | 1 | 0
Period: OLE Phase (48 Weeks)
Arm/Group | Verdiperstat | Placebo
Started | 123 (Participants who continued into the extension phase.) | 140 (Participants who continued into the extension phase.)
Completed | 44 | 46
Not Completed | 79 | 94
Not completed — Adverse Event | 18 | 29
Not completed — Disease Progression | 6 | 9
Not completed — Participant Request to Discontinue | 35 | 38
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Other | 16 | 13

BASELINE CHARACTERISTICS:
Population: Treated participants included enrolled participants who received at least 1 dose of blinded study therapy (verdiperstat or placebo).
Groups:
- Verdiperstat: Randomization phase (Randomization through Week 48): Participants received verdiperstat 300 mg tablet orally once daily for 1 week, followed by 300 mg twice daily for 1 week, and then 600 mg twice daily for the remaining 46 weeks of the double-blind phase.
  OLE phase (48 weeks): Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to continue verdiperstat 600 mg orally twice daily for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Verdiperstat | Placebo | Total
Number analyzed (Participants) | 168 | 168 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (7.12) | 60.1 (6.68) | 61.3 (6.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 83 | 166
  Male | 85 | 85 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 163 | 163 | 326
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  White | 155 | 156 | 311
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Unified Multiple System Atrophy Rating Scale (UMSARS) Modified Score [Mean (Standard Deviation); unit: units on a scale] — UMSARS - clinician-rated scale comprised of 4 parts: Part I (Historical Review), Part II (Motor Examination), Part III (Autonomic Examination), Part IV (Global Disability Scale). Modified UMSARS is composed of subset of 9 items from original UMSARS Part I and Part II. Responses are measured on 4-point scale ranged from 0-3. Total modified UMSARS score is sum of these 9 items, score range from 0 to 27. Higher scores indicate greater impairment.
  units on a scale | 6.1 (4.24) | 5.8 (3.74) | 6.0 (3.99)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Modified UMSARS Score at Week 48
Description: UMSARS - clinician-rated scale comprised of 4 parts: Part I (Historical Review), Part II (Motor Examination), Part III (Autonomic Examination), Part IV (Global Disability Scale). Modified UMSARS is composed of subset of 9 items from original UMSARS Part I and Part II. Responses are measured on 4-point scale ranged from 0-3, where 0= no/mild impairment, 1= moderate impairment, 2= severe impairment, 3=complete impairment. Total modified UMSARS score is sum of these 9 items, score range from 0 to 27. Higher scores indicate greater impairment.
Time Frame: Baseline and Week 48
Population: Modified Intent to Treat (mITT) population included randomized participants who received at least 1 dose of blinded study therapy and provided a baseline and at least 1 post-baseline efficacy assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Verdiperstat - Randomization Phase: Randomization phase (Randomization through Week 48): Participants received verdiperstat 300 mg tablet orally once daily for 1 week, followed by 300 mg twice daily for 1 week, and then 600 mg twice daily for the remaining 46 weeks of the double-blind phase.
- Placebo - Randomization Phase: Randomization phase (Randomization through Week 48): Participants received placebo matching with verdiperstat for 48 weeks.
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 125 | 140
units on a scale | 5.20 [4.52 to 5.89] | 4.85 [4.19 to 5.51]
Statistical Analysis 1: Comparison: Verdiperstat - Randomization Phase vs Placebo - Randomization Phase; Test type: Superiority; p = 0.4656, Mixed Models Analysis; Least Square mean difference = 0.35, 95% CI 2-sided [-0.60 to 1.30], Standard Error of Mean 0.48

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in participants or clinical investigation participants administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. A serious AE (SAE) is defined as any event that met any of the following criteria at any dose: death; life-threatening; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect in the offspring of a participant who received study drug; other important medical events that may not have resulted in death, be life-threatening, or required hospitalization, or, based upon appropriate medical judgment, they may have jeopardized the participant and may have required medical or surgical intervention to prevent one of the other serious outcomes.
Time Frame: Up to 100 weeks
Population: Treated population included enrolled participants who received at least 1 dose of blinded study therapy (verdiperstat or placebo).
Measure: Number; unit: participants
Groups:
- Verdiperstat - Randomization Phase: Participants received verdiperstat 300 mg tablet orally once daily for 1 week, followed by 300 mg twice daily for 1 week, and then 600 mg twice daily for the remaining 46 weeks of the double-blind phase.
- Placebo - Randomization Phase: Participants received placebo matching with verdiperstat for 48 weeks.
- Verdiperstat - Randomization Phase/ Verdiperstat - OLE Phase: Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to continue verdiperstat 600 mg orally twice daily for 48 weeks.
- Placebo - Randomization Phase/ Verdiperstat - OLE Phase: Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to receive verdiperstat 600 mg tablet orally twice daily for 48 weeks.
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase | Verdiperstat - Randomization Phase/ Verdiperstat - OLE Phase | Placebo - Randomization Phase/ Verdiperstat - OLE Phase
Number analyzed (Participants) | 168 | 168 | 123 | 140
participants
  TEAE | 160 | 156 | 95 | 112
  Serious TEAE | 44 | 29 | 30 | 27

3. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Week 48
Description: The CGI-I is a clinician-rated scale measuring the change in the participant's clinical status from a specific point in time. It is scored on a 7- point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change. Higher scores indicate greater impairment.
Time Frame: Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 126 | 142
units on a scale | 5.07 [4.92 to 5.21] | 5.14 [5.00 to 5.27]

4. Secondary Outcome: Change From Baseline in Multiple System Atrophy Quality of Life (MSA-QoL) Motor Subscale at Week 48
Description: The MSA-QoL is a participant-rated scale that was designed to measure health-related quality of life specifically in MSA. It assesses activities of daily living and has subscales for motor, nonmotor, and emotional/social domains. The MSA-QoL motor subscale includes 14 items. The response to each question ranges from 0= no problem, to 4= extreme problem, with a total scale ranging from 0-56. Higher scores indicates higher impact of the disease on the aspect measured by each subscale.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 114 | 130
units on a scale | 13.83 [10.97 to 16.69] | 13.45 [10.72 to 16.18]

5. Secondary Outcome: Change From Baseline in Multiple System Atrophy Quality of Life (MSA-QoL) Non-motor Subscale at Week 48
Description: The MSA-QoL is a participant-rated scale that was designed to measure health-related quality of life specifically in MSA. It assesses activities of daily living and has subscales for motor, nonmotor, and emotional/social domains. The MSA-QoL nonmotor subscale includes 12 items. The response to each question ranges from 0= no problem, to 4= extreme problem, with a total scale ranging from 0-48. Higher scores indicates higher impact of the disease on the aspect measured by each subscale.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 116 | 128
units on a scale | 7.52 [4.93 to 10.11] | 5.56 [3.07 to 8.04]

6. Secondary Outcome: Change From Baseline in UMSARS Part I and Part II Total Score at Week 48
Description: The UMSARS is a clinician-rated scale comprised of 4 parts: Part I (Historical Review with 12 questions), Part II (Motor Examination with 14 questions), Part III (Autonomic Examination), and Part IV (Global Disability Scale). UMSARS Part I and Part II responses are measured on a 5-point scale ranging from 0 to 4, where 0= no impairment, 1= mild impairment, 2= moderate impairment, 3= severe impairment, 4=complete impairment. Each subscale score is a sum of its items and total score is sum of all 26 items, score range from 0 to 104. Higher scores indicates greater impairment.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 125 | 139
units on a scale | 12.00 [10.37 to 13.63] | 11.34 [9.77 to 12.90]

7. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S) at Week 48
Description: The PGI-S is a participant-rated scale that measures how participants perceive the severity of their illness. The PGI-S is a 1-item questionnaire on a 4-point scale ranging from 1 to 4, where, 1 = normal, 2 = mild, 3 = moderate, 4 = severe. Higher scores indicate greater impairment.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 125 | 142
units on a scale | 0.33 [0.23 to 0.42] | 0.27 [0.18 to 0.36]

8. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) at Week 48
Description: The CGI-S is a clinician-rated scale measuring the severity of the participant's illness. It is scored on a 7- point scale ranging from 1 (normal, not ill at all) to 7 (among the most extremely ill patients). Higher scores indicate greater impairment.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 126 | 142
units on a scale | 0.79 [0.66 to 0.92] | 0.78 [0.66 to 0.90]

9. Secondary Outcome: Change From Baseline in UMSARS Part III at Week 48 (Blood Pressure (BP) Only)
Description: The UMSARS is a clinician-rated scale comprised of 4 parts: Part I (Historical Review), Part II (Motor Examination), Part III (Autonomic Examination) and Part IV (Global Disability Scale). Only Part III of UMSARS was analyzed. Part III of the UMSARS is an Autonomic Exam, consisting of Supine and Standing Systolic and Diastolic Blood Pressure, Heart rate and presence Orthostatic Symptoms. Only change in Orthostatic Blood Pressure reported.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter of mercury
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 118 | 132
millimeter of mercury
  Change in Orthostatic Systolic BP | -2.18 [-5.90 to 1.55] | -3.09 [-6.63 to 0.44]
  Change in Orthostatic Diastolic BP: number analyzed (Participants) | 118 | 131
  Change in Orthostatic Diastolic BP | -2.87 [-5.13 to -0.61] | -2.54 [-4.70 to -0.38]

10. Secondary Outcome: Change From Baseline in UMSARS Part III at Week 48 (Heart Rate (HR) Only)
Description: The UMSARS is a clinician-rated scale comprised of 4 parts: Part I (Historical Review), Part II (Motor Examination), Part III (Autonomic Examination) and Part IV (Global Disability Scale). Only Part III of UMSARS was analyzed. Part III of the UMSARS is an Autonomic Exam, consisting of Supine and Standing Systolic and Diastolic Blood Pressure, Heart rate and presence Orthostatic Symptoms. Only change in Orthostatic Heart Rate reported.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 119 | 132
beats per minute | 0.20 [-1.48 to 1.87] | -0.68 [-2.27 to 0.91]

11. Secondary Outcome: Change From Baseline in UMSARS Part IV at Week 48
Description: The UMSARS is a clinician-rated scale comprised of 4 parts: Part I (Historical Review), Part II (Motor Examination), Part III (Autonomic Examination) and Part IV (Global Disability Scale). Only Part IV of UMSARS was analyzed. Part IV was measured on a 5-point scale ranging from 1= Completely independent. Able to do all chores with minimal difficulty or impairment. Essentially normal. Unaware of any difficulty, to 5= Totally dependent and helpless. Bedridden. Higher scores indicate greater impairment.
Time Frame: Baseline and Week 48
Population: mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase
Number analyzed (Participants) | 126 | 140
units on a scale | 0.82 [0.69 to 0.96] | 0.85 [0.72 to 0.99]

ADVERSE EVENTS:
Time Frame: TEAEs were reported from first dose of study drug and prior to 30 days after the last dose of study drug, maximum of 100 weeks.
Description: Treated population included enrolled participants who received at least 1 dose of blinded study therapy (verdiperstat or placebo).
Groups:
- Verdiperstat - Randomization Phase/Verdiperstat - OLE Phase: Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to continue verdiperstat 600 mg orally twice daily for 48 weeks.
- Placebo - Randomization Phase/Verdiperstat - OLE Phase: Participants who completed the double-blind phase were offered the opportunity to enroll in an OLE phase to receive verdiperstat 600 mg tablet orally twice daily for 48 weeks.
Arm/Group | Verdiperstat - Randomization Phase | Placebo - Randomization Phase | Verdiperstat - Randomization Phase/Verdiperstat - OLE Phase | Placebo - Randomization Phase/Verdiperstat - OLE Phase
All-Cause Mortality (participants affected / at risk) | 11/168 | 5/168 | 12/123 | 10/140
Serious Adverse Events (participants affected / at risk) | 44/168 | 29/168 | 30/123 | 27/140
Other Adverse Events (participants affected / at risk) | 125/168 | 130/168 | 55/123 | 71/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verdiperstat - Randomization Phase (N=168) | Placebo - Randomization Phase (N=168) | Verdiperstat - Randomization Phase/Verdiperstat - OLE Phase (N=123) | Placebo - Randomization Phase/Verdiperstat - OLE Phase (N=140)
Urinary tract infection (Infections and infestations) | 7 (11) | 1 (1) | 4 (4) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2) | 1 (2) | 1 (1)
Urosepsis (Infections and infestations) | 4 (4) | 2 (3) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 2 (4) | 1 (1) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bradykinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Pericarditis constrictive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dorsal ramus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verdiperstat - Randomization Phase (N=168) | Placebo - Randomization Phase (N=168) | Verdiperstat - Randomization Phase/Verdiperstat - OLE Phase (N=123) | Placebo - Randomization Phase/Verdiperstat - OLE Phase (N=140)
Urinary tract infection (Infections and infestations) | 44 (71) | 54 (77) | 26 (38) | 29 (40)
COVID-19 (Infections and infestations) | 2 (2) | 11 (11) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 21 (25) | 23 (28) | 3 (4) | 11 (12)
Dizziness (Nervous system disorders) | 13 (16) | 22 (22) | 3 (3) | 5 (6)
Balance disorder (Nervous system disorders) | 17 (20) | 14 (15) | 3 (4) | 4 (5)
Syncope (Nervous system disorders) | 3 (4) | 9 (11) | 2 (5) | 8 (8)
Fall (Injury, poisoning and procedural complications) | 37 (66) | 39 (53) | 21 (27) | 21 (38)
Fatigue (General disorders) | 15 (15) | 14 (17) | 6 (6) | 4 (4)
Gait disturbance (General disorders) | 12 (12) | 12 (12) | 2 (2) | 2 (2)
Oedema peripheral (General disorders) | 12 (12) | 7 (8) | 6 (6) | 4 (4)
Constipation (Gastrointestinal disorders) | 19 (21) | 12 (13) | 7 (7) | 4 (6)
Nausea (Gastrointestinal disorders) | 17 (19) | 8 (8) | 1 (1) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 9 (10) | 3 (3) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 3 (3) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 7 (7) | 11 (12) | 4 (4) | 4 (4)
Hypertension (Vascular disorders) | 3 (3) | 9 (9) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 10 (11) | 7 (7) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 9 (12) | 4 (5) | 1 (1) | 4 (5)
Blood thyroid stimulating hormone increased (Investigations) | 9 (13) | 1 (1) | 6 (6) | 7 (7)
Asthenia (General disorders) | 7 (7) | 6 (7) | 5 (5) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/06/NCT03952806/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03952806/SAP_001.pdf